CLINICAL TRIAL: NCT02636504
Title: Evaluation of Three Pulp Vitality Tests
Status: Not yet recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAO5900
Record Dates: First submitted 2015-12-16; First posted 2015-12-21 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Dental Pulp Diseases; Dental Pulp Vitality Testing
Keywords: Pulp vitality; Pulp testing
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Laser-Doppler Flowmetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Laser Doppler Flowmetry — Pulp vitality of teeth is tested with three pulp vitality testing including laser Doppler flowmetry, cold testing, and electric pulp testing.
  Other Names: Cold testing; Electric Pulp Testing

SUMMARY:
The objectives of this study are to determine the sensitivity, specificity, positive predictive value, negative predictive value, and accuracy of laser Doppler flowmetry in determining the vitality of teeth and comparing with those of electric pulp testing and cold testing.

DETAILED DESCRIPTION:
Prior to starting any endodontic treatment, it is essential to determine the vitality of the tooth in question. Vitality of a tooth is defined as the presence of blood flow into the tooth. The vitality status of a tooth will affect the success of endodontic treatment, and therefore plays an important role in treatment planning. Two established methods of determining vitality are electric pulp tests and cold tests. However, both these methods have drawbacks. Both methods use the presence of sensory feedback in the tooth as a predictor of tooth vitality. This can lead to errors because blood flow and nerves in the tooth may be lost at different times, resulting in false-positive and false-negative responses. Both are subjective and patient-dependent, relying on the patient to indicate when pain is felt. In addition, studies have suggested that electric pulp testing and cold tests are not as reliable in immature teeth, teeth undergoing orthodontic movement, traumatized teeth, and teeth with significant secondary dentin. Laser Doppler flowmetry is a technique that utilizes the Doppler principle to determine blood flow. It has been used widely in the medical field to measure blood flow in the skin. Some studies have also shown good results in measuring blood flow in the pulp of teeth. The objectives of this study are to determine the sensitivity, specificity, positive predictive value, negative predictive value, and accuracy of laser Doppler flowmetry in determining the vitality of teeth and comparing with those of electric pulp testing and cold testing.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for inclusion in the study will be that the individual has teeth that require endodontic treatment and patient is willing to undergo two additional vitality tests which will take about 20 minutes of additional time.

Exclusion Criteria:

* No group of special subjects or vulnerable population is being targeted in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that need endodontic treatment will have a consultation visit first. In most cases, the endodontic treatment will be provided at a subsequent visit. In some cases the endodontic treatment will be provided at the same visit. Patients who present to the endodontic clinic for a consultation visit for endodontic treatment. The patient will have three types of pulp vitality tests done on the tooth that is to receive endodontic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The number of teeth showing the true positive, true negative, false positive, and false negative after pulp vitality testing | 1 year
  Patients who present to the endodontic clinic for a consultation visit prior to treatment. The patient will have three types of pulp vitality tests done on the tooth that is to receive endodontic treatment. The number of teeth that show the true positive, true negative, false positive, and false negative after pulp vitality testing will be measured. For example, a tooth that is diagnosed nonvital based on the pulp vitality testing will be confirmed when endodontic treatment is performed. If there is a discrepancy, it can be counted as false negative. When a tooth is diagnosed vital based on the pulp testing and confirmed to be vital, it can be counted as true positive. When a tooth is diagnosed vital based on the pulp testing and confirmed to be nonvital, it can be counted as false positive. When a tooth is diagnosed nonvital and confirmed novital, it is counted as true negative.

CONTACTS AND LOCATIONS:
Overall Officials: Sahng G Kim, DDS, MS, Principal Investigator — Columbia University College of Dental Medicine
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Karayilmaz H, Kirzioglu Z. Comparison of the reliability of laser Doppler flowmetry, pulse oximetry and electric pulp tester in assessing the pulp vitality of human teeth. J Oral Rehabil. 2011 May;38(5):340-7. doi: 10.1111/j.1365-2842.2010.02160.x. Epub 2010 Sep 26. PMID 20868433
- [Background] Chen E, Abbott PV. Evaluation of accuracy, reliability, and repeatability of five dental pulp tests. J Endod. 2011 Dec;37(12):1619-23. doi: 10.1016/j.joen.2011.07.004. Epub 2011 Sep 9. PMID 22099893